CLINICAL TRIAL: NCT07094477
Title: An Exploratory Clinical Study on Targeted CD22/CD19 CAR-T Cell Immunotherapy for First-line Consolidation Therapy of High-risk Invasive B-cell Lymphoma
Brief Title: Study of Targeted CD22/CD19 CAR-T Therapy for First-line Consolidation of B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daihong Liu (Other)
Responsible Party: Sponsor-Investigator, Daihong Liu, Dr., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-124-01
Record Dates: First submitted 2025-06-01; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma
Keywords: B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Prospective Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): patients with high-risk invasive B-cell lymphoma who accept targeted CD22/CD19 CAR-T cell immunotherapy for first-line consolidation therapy
  Interventions: Drug: CD22/CD19 CAR-T cell immunotherapy

INTERVENTIONS:
Drug: CD22/CD19 CAR-T cell immunotherapy — targeted CD22/CD19 CAR-T cell immunotherapy
  Other Names: CAR-T cell immunotherapy

SUMMARY:
The purpose of this study is to determine the efficacy and safety of targeted CD22/CD19 CAR-T cell immunotherapy for first-line consolidation therapy of high-risk invasive B-cell lymphoma.

DETAILED DESCRIPTION:
Only a portion of patients with invasive B-cell lymphoma can achieve complete response through standard combination therapy with R-CHOP, and a considerable number of patients have poor prognosis and face treatment difficulties such as drug resistance and recurrence.

In the previous guidelines of the National Comprehensive Cancer Network (NCCN) in the United States, high-risk diffuse large B-cell lymphoma (defined as stage III-IV, or stage I-II with extensive mesenteric involvement) patients showed complete response after completing six cycles of first-line induction therapy. Subsequently, autologous stem cell transplantation (ASCT) and involved site radiation therapy (ISRT) can be used for consolidation treatment. However, the SWOG 9704 study found that patients with medium to high risk/high-risk B-cell lymphoma who achieved at least partial response to first-line treatment and received ASCT consolidation therapy did not benefit from ASCT in terms of progression free survival/overall survival in the medium to high risk group, only in terms of overall survival and disease-free survival in the high-risk group. In addition, the DLCL04 study showed that medium to high-risk or high-risk patients with an Age Adjusted International Prognostic Index (aaIPI) score of 2-3 who achieved complete or partial response to first-line treatment did not benefit from ASCT.

In the 2024 NCCN guidelines for diffuse large B-cell lymphoma, first-line consolidation therapy for high-risk diffuse large B-cell lymphoma patients after induction therapy only includes close follow-up and radiation consolidation therapy for the affected areas of the original mass and bone lesions. There is no more aggressive treatment strategy to positively address the relatively high risk of disease recurrence and progression in this group of high-risk patients.

CAR-T cell immunotherapy has achieved good clinical therapeutic effects in hematological tumors. After induction therapy, first-line CAR-T cell immunotherapy consolidation therapy is expected to improve the disease prognosis of high-risk invasive B-cell lymphoma patients and bring long-term survival benefits. Compared to CAR-T cell immunotherapy, which can directly control adverse reactions with immunosuppressive drugs such as glucocorticoids, the risk of autologous hematopoietic stem cell transplantation is higher, and patients have a greater risk of non recurrent mortality (NRM) due to complications such as infection and bleeding. The latest version of the NCCN guidelines for diffuse large B-cell lymphoma no longer recommends autologous hematopoietic stem cell transplantation as the first-line consolidation treatment for high-risk diffuse large B-cell lymphoma. Therefore, new first-line consolidation treatment plans after induction therapy are still needed to further improve the survival prognosis of high-risk invasive B-cell lymphoma patients.

Based on the many difficulties that still exist in the first-line standard treatment plan for high-risk invasive B-cell lymphoma patients, this study plans to explore the effectiveness and safety of CD22/CD19 CAR-T cell immunotherapy as first-line consolidation therapy for high-risk invasive B-cell lymphoma patients after standard first-line induction therapy, in order to improve the prognosis of such patients and provide new treatment options for first-line consolidation therapy of high-risk invasive B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. With the patient's consent and signed informed consent form, willing and able to comply with the planned visits, research treatments, laboratory tests, and other experimental procedures; 2. CD19 and/or CD22 positive large B-cell lymphoma (LBCL) diagnosed by cytology or histology according to WHO 2016 standards, including diffuse large B-cell lymphoma (DLBCL), high-grade lymphoma (HGBL), etc.: 1) The patient's disease is still evaluated as partial response (PR) after induction treatment with standard first-line chemotherapy regimen, or 2) The patient's disease reaches complete response (CR) after induction treatment with standard first-line chemotherapy regimen, but there are high-risk factors at the time of onset; 3. The possible high-risk factors for the patient's onset of the disease are as follows: 1) FISH confirmed high-grade B-cell lymphoma with double or triple strikes, accompanied by MYC and BCL2 and/or BCL6 rearrangements; 2) Advanced B-cell lymphoma with 11q abnormalities/Burkitt like lymphoma with 11q abnormalities; 3) The International Prognostic Index (IPI) at the time of initial diagnosis is 2-5 points; The Age Adjusted International Prognostic Index (aaIPI) is 2-3 points; The National Comprehensive Cancer Network International Prognostic Index (NCCN-IPI) score ranges from 4-8 points in the United States; 4) Immunohistochemical CD5 positivity; 5) Immunohistochemistry suggests dual expression of MYC and BCL-2 (recommended dual expression threshold is MYC ≥ 40%, BCL2 ≥ 50%); 6) Gene sequencing shows TP53 mutation; 7) The second-generation sequencing (NGS) suggests molecular typing as MCD subtype and N1 subtype; 4. Age range from 18 to 85 years old, male or female; 5. Subjects with physical fitness status scores ranging from 0 to 2 in the Eastern Cooperative Oncology Group (ECOG) in the United States; 6. Expected survival period from the date of signing the informed consent form is greater than 3 months; 7. HGB ≥ 60g/L; 8. The absolute value of neutrophils in peripheral blood is ≥ 1000/μl, and the platelet count is ≥ 45000/μl; 9. Liver and kidney function, as well as heart and lung function, meet the following requirements: 1) Total bilirubin (TBIL) ≤ 1.5 times the upper limits of normal (ULN), except for subjects with Gilbert's syndrome; 2) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN; 3) Serum Creatinine (Cr) ≤ 1.5 times ULN or Creatinine Clearance Rate (CCr) ≥ 60mL/min, estimated based on the Cockcroft Gault formula; 4) The left ventricular ejection fraction (LVEF) of the heart is ≥ 50%. Echocardiography (ECHO) confirms no pericardial effusion and no clinically significant arrhythmia; 5) Baseline transcutaneous oxygen saturation under indoor ventilation>92%; 6) No clinically significant pleural effusion; 10. Participants with pregnancy plans must agree to take contraceptive measures for a continuous period of 6 months from before enrollment in the study until the end of the study; If the subject is pregnant or suspected of being pregnant, the researcher should be notified immediately.

Exclusion Criteria:

* 1. Have received any form of chimeric antigen receptor cell therapy or other genetically modified T cell therapy; 2. Has a history of severe immediate hypersensitivity reactions to aminoglycoside antibiotics and other essential medications; 3. Known history of human immunodeficiency virus (HIV) infection or active hepatitis B virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotics (active HBV infection is defined as: a. HBV DNA quantification ≥ 2000 IU/ml; b. ALT ≥ 2 times the normal upper limit value; c. Exclude hepatitis caused by the disease itself, medication, or other reasons; All three conditions must be met simultaneously. If a patient is diagnosed with active HBV infection at the time of initial diagnosis and becomes non active HBV infection after anti HBV treatment, they can be included in this study under the premise of sufficient anti HBV treatment; 4. Non hematological tumors (such as lymphoma) associated liver and kidney dysfunction: ALT>3 times the upper limit of normal, AST>3 times the upper limit of normal, TBIL>2 times the upper limit of normal, serum creatinine clearance rate<30 mL/min; 5. History of myocardial infarction, cardiac angioplasty or coronary stent implantation, unstable angina, active arrhythmia, or other clinically significant cardiovascular diseases within the 12 months prior to enrollment; 6. Other serious medical diseases may have an impact on this study (such as diabetes, gastric ulcer, other serious respiratory and circulatory diseases, severe autoimmune diseases or congenital immune defects, severe infection and inability to be effectively controlled), as well as other diseases with high risk of disease change; 7. Has a history of severe immediate hypersensitivity reactions to any medication necessary for use in this study; History of severe allergy to biological products (including antibiotics); 8. Female subjects who are currently pregnant or breastfeeding (with potential risks to the fetus or infant from pre-treatment chemotherapy regimens); 9. The researchers determined that the subjects were unable to complete all the required visit surveys or diagnostic procedures (including medium - and long-term follow-up visits) as per the study protocol, had poor willingness to participate in the study, were unwilling to join and fully comply with the study arrangements, and had insufficient compliance with the study by the subjects and their families. The decision-making power belongs to the researcher; 10. The subjects who have previously suffered from other malignant tumors cannot be included in this study unless they are disease-free and have not received any form of anti-tumor treatment for at least 3 years (except for skin tumors of non malignant melanoma and in situ cancers occurring in the cervix, bladder, breast, etc.); 11. History of receiving live vaccines within 6 weeks prior to initiating the pre-treatment plan; 12. Those who have undergone large-scale surgical treatment (excluding lymph node biopsy) within the past 14 days, or those who are expected to undergo large-scale surgical treatment during the treatment process; 13. There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, or interfere with the study results, as well as patients deemed unsuitable by the researchers to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
1-year progression free survival rate (1-year-PFS) | 1 year after treatment
  The 1-year progression free survival rate (1-year-PFS) of targeted CD22/CD19 CAR-T cell immunotherapy for first-line consolidation therapy of high-risk invasive B-cell lymphoma refers to the proportion of disease progression that occurs within one year after treatment in patients.

SECONDARY OUTCOMES:
overall survival (OS) | 1 year after treatment
  Overall survival (OS) refers to the time from the start of treatment to the death of the patient for any reason.
time to progression (TTP) | 1 year after treatment
  Time to progression (TTP) refers to the time from treatment to the first lymphoma progression.
disease free survival (DFS) | 1 year after treatment
  Disease free survival (DFS) refers to the time from treatment to the first lymphoma recurrence.
duration of response (DOR) | 1 year after treatment
  Duration of Response (DOR) refers to the time from the first assessment of a lymphoma as a complete or partial response to the first assessment of PD (Progressive Disease) or death from any cause.
event free survival (EFS) | 1 year after treatment
  Event Free Survival (EFS) is a commonly used endpoint indicator in clinical trials to evaluate the survival time of patients without any adverse events during a specific time period. These adverse events include but are not limited to disease progression, death, treatment plan changes, and the occurrence of serious side effects.
recurrence rate | 1 year after treatment
  The recurrence rate refers to the proportion of patients with lymphoma recurrence after treatment.
Treatment-related safety indicators | 1 year after treatment
  The safety of this CD22/CD19 CAR-T cell immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-Hong Liu, Dr., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive personal health information

REFERENCES:
- [Background] Khan AN, Asija S, Pendhari J, Purwar R. CAR-T cell therapy in hematological malignancies: Where are we now and where are we heading for? Eur J Haematol. 2024 Jan;112(1):6-18. doi: 10.1111/ejh.14076. Epub 2023 Aug 7. PMID 37545253
- [Background] Baker DJ, Arany Z, Baur JA, Epstein JA, June CH. CAR T therapy beyond cancer: the evolution of a living drug. Nature. 2023 Jul;619(7971):707-715. doi: 10.1038/s41586-023-06243-w. Epub 2023 Jul 26. PMID 37495877
- [Background] CD19/CD22 Dual-Targeted CAR-T Therapy Active in Relapsed/Refractory DLBCL. Oncologist. 2020 Jul;25 Suppl 1(Suppl 1):S12-S13. doi: 10.1634/theoncologist.2020-0560. Epub 2020 Jun 26. PMID 32589304
- [Background] Nguyen TT, Thanh Nhu N, Chen CL, Lin CF. Effectiveness and safety of CD22 and CD19 dual-targeting chimeric antigen receptor T-cell therapy in patients with relapsed or refractory B-cell malignancies: A meta-analysis. Cancer Med. 2023 Sep;12(18):18767-18785. doi: 10.1002/cam4.6497. Epub 2023 Sep 5. PMID 37667978
- [Background] Zeng C, Cheng J, Li T, Huang J, Li C, Jiang L, Wang J, Chen L, Mao X, Zhu L, Lou Y, Zhou J, Zhou X. Efficacy and toxicity for CD22/CD19 chimeric antigen receptor T-cell therapy in patients with relapsed/refractory aggressive B-cell lymphoma involving the gastrointestinal tract. Cytotherapy. 2020 Mar;22(3):166-171. doi: 10.1016/j.jcyt.2020.01.008. Epub 2020 Feb 13. PMID 32063474
- [Background] Spiegel JY, Patel S, Muffly L, Hossain NM, Oak J, Baird JH, Frank MJ, Shiraz P, Sahaf B, Craig J, Iglesias M, Younes S, Natkunam Y, Ozawa MG, Yang E, Tamaresis J, Chinnasamy H, Ehlinger Z, Reynolds W, Lynn R, Rotiroti MC, Gkitsas N, Arai S, Johnston L, Lowsky R, Majzner RG, Meyer E, Negrin RS, Rezvani AR, Sidana S, Shizuru J, Weng WK, Mullins C, Jacob A, Kirsch I, Bazzano M, Zhou J, Mackay S, Bornheimer SJ, Schultz L, Ramakrishna S, Davis KL, Kong KA, Shah NN, Qin H, Fry T, Feldman S, Mackall CL, Miklos DB. CAR T cells with dual targeting of CD19 and CD22 in adult patients with recurrent or refractory B cell malignancies: a phase 1 trial. Nat Med. 2021 Aug;27(8):1419-1431. doi: 10.1038/s41591-021-01436-0. Epub 2021 Jul 26. PMID 34312556
- [Background] Wei G, Zhang Y, Zhao H, Wang Y, Liu Y, Liang B, Wang X, Xu H, Cui J, Wu W, Zhao K, Nagler A, Chang AH, Hu Y, Huang H. CD19/CD22 Dual-Targeted CAR T-cell Therapy for Relapsed/Refractory Aggressive B-cell Lymphoma: A Safety and Efficacy Study. Cancer Immunol Res. 2021 Sep;9(9):1061-1070. doi: 10.1158/2326-6066.CIR-20-0675. Epub 2021 Jul 21. PMID 34290048